CLINICAL TRIAL: NCT03905564
Title: Single Site, Open-label, Randomized, Two Treatments, Two Periods, Two Sequences, Crossover Trial to Evaluate the Bioequivalence of Two Delayed-release Oral Formulations of a Fixed Combination of Doxylamine Succinate 10 mg/Pyridoxine Hydrochloride 10 mg (Test Product: Product of Tecnandina, S.A. TENSA; Reference Product: Diclegis (Registered Trademark) Product of Duchesnay Inc.) After a Single Administration of Two Tablets to Healthy Women Under Fasting Conditions
Brief Title: A Study to Investigate Differences in the Extent and Rate of Absorption of Doxylamine/Pyridoxine From 2 Different Products Under Fasting Conditions
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Grünenthal, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP8012-01; DXLPRD-06-GRU (Other: Sponsor code); 17-CI-09 012 084 (Registry Identifier: COFEPRIS (Comisión Federal para la Protección contra Riesgos Sanitarios))
Record Dates: First submitted 2019-02-20; First posted 2019-04-05 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Bioavailability
MeSH Terms: interventions — doxylamine succinate; Pyridoxine; dicyclomine, doxylamine, pyridoxine drug combination

STUDY DESIGN:
Intervention Model Description: Randomized, single-dose with two periods, two sequences (AB, BA; A = Reference and B = Test) crossover study in healthy participants under fasting conditions. Washout period between the two study periods will be at least 20 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxylamine succinate/pyridoxine hydrochloride (Experimental): Oral single dose equivalent to doxylamine succinate 20 mg and pyridoxine hydrochloride 20 mg (i.e., 2 tablets doxylamine succinate 10 mg/pyridoxine hydrochloride 10 mg combination) administered with 250 mL of water (at room temperature) under fasting conditions.
  Interventions: Drug: doxylamine succinate 10 mg/pyridoxine hydrochloride 10 mg combination
- Diclegis (Registered Trademark) (Active Comparator): Oral single dose equivalent to doxylamine succinate 20 mg and pyridoxine hydrochloride 20 mg (i.e., 2 tablets) administered with 250 mL of water (at room temperature) under fasting conditions.
  Interventions: Drug: Diclegis (Registered Trademark)

INTERVENTIONS:
Drug: doxylamine succinate 10 mg/pyridoxine hydrochloride 10 mg combination — Delayed-release tablet containing a fixed-dose combination of doxylamine succinate 10 mg and pyridoxine hydrochloride 10 mg (product of Tecnandina, S.A. TENSA).
  Arms: Doxylamine succinate/pyridoxine hydrochloride
Drug: Diclegis (Registered Trademark) — Delayed-release tablet containing a fixed-dose combination of doxylamine succinate 10 mg and pyridoxine hydrochloride 10 mg (product of Duchesnay Inc.).
  Arms: Diclegis (Registered Trademark)

SUMMARY:
The purpose of the study is to investigate any difference in the extent and rate of absorption of doxylamine between the test (investigational medicinal product [IMP]) and reference products that could impact the bioavailability of the medication when administered under fasting conditions.

DETAILED DESCRIPTION:
The objective of the study is to compare the bioavailability of doxylamine between two oral delayed-release formulations containing the fixed-dose combination of doxylamine succinate 10 milligrams (mg)/pyridoxine hydrochloride 10 mg

* A product of Tecnandina, S.A. TENSA (Test) and
* Diclegis (Registered Trademark), a product of Duchesnay Inc.(Reference)

after an administration of a single dose equivalent to doxylamine succinate 20 mg and pyridoxine hydrochloride 20 mg (i.e., 2 tablets) under fasting conditions to determine bioequivalence in terms of rate and extent of absorption.

Furthermore, the tolerability of the fixed-dose combination doxylamine succinate 10 mg/pyridoxine hydrochloride 10 mg will be evaluated in healthy women in a dose equivalent to doxylamine succinate 20 mg and pyridoxine hydrochloride 20 mg.

ELIGIBILITY:
Inclusion Criteria:

* Participation will be voluntary and according to the guidelines proposed by the Health General Law and informed consent will be obtained according to the previously mentioned law. In addition, the study will be conducted according to the ethical principles that have their origin in the Declaration of Helsinki, the review of Brazilian laws, and Good Clinical Practice.
* Only healthy female participants aged between 18 and 55 years will be included.
* The body mass index must be between 18.0 and 27.0 kilograms per square meter according to the Quetelet index.
* Participants must be willing to use contraceptive methods (including barrier methods, non-hormonal intra-uterine device, or have a preexistent bilateral tubal ligation) during the conduct of the study and for up to 3 weeks after the last dose is administered.
* Participants must be healthy as determined by the results of a complete clinical history recorded by the clinical investigational site physicians and the results of the laboratory examinations and 12-lead electrocardiogram done by a certified clinical laboratory.
* The allowed limits of variation within normal in the screening visit will be: systolic blood pressure (sitting) less or equal to 120 mmHg, diastolic blood pressure less or equal to 80 mm Hg, heart rate between 50 and 100 beats per minute and respiratory rate between 14 and 20 breaths per minute according to the current standard operating procedure. Vital signs will be measured after 10 minutes of resting in a sitting position.
* Laboratory and other examinations to be conducted for the inclusion of participants will be:

  1. Complete blood count: leukocytes, erythrocytes, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, erythrocyte distribution width, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils.
  2. Blood chemistry 27 elements: glucose, urea, blood urea nitrogen (BUN), creatinine, BUN/creatinine ratio, uric acid, cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides, low-density lipoprotein cholesterol, non-HDL cholesterol, atherogenic index, total protein, albumin, globulins, albumin/globulin ratio, total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, total alkaline phosphatase, gamma-glutamyl transferase, lactate dehydrogenase, iron, calcium, sodium, potassium, and chloride.
  3. Urinalysis: Physical examination (color, appearance, density); chemical examination (pH, leukocytes, nitrite, protein, glucose, ketones, bilirubin, urobilinogen, hemoglobin); microscopic examination (leukocytes, erythrocytes, dysmorphic erythrocytes, casts, crystals, squamous epithelial cells, tubular renal cells, mucus, bacteria and yeasts).
  4. Hepatitis B screening (Anti-HBc = Antibody to hepatitis B core antigen, HBs-Ab = antibody to hepatitis B surface antigen, Anti-HBs = antibody to hepatitis B surface antigen) and hepatitis C antibodies.
  5. HIV test: Antibodies to the human immunodeficiency virus (Anti-HIV 1 and 2).
  6. Venereal disease research laboratory (VDRL) test.
  7. Urine drugs of abuse test at the screening visit and at approximately 12 hours prior to the administration of the IMP in both study periods.
  8. Alcohol breath test approximately 12 hours prior to the administration of the IMP in both study periods.
  9. Serum pregnancy test (beta-human chorionic gonadotropin) at the screening visit and urine pregnancy test (qualitative) at approximately 12 hours prior to the administration of the IMP in both study periods.
  10. 12-lead electrocardiogram which will be performed after resting for 10 minutes in a sitting position.

Exclusion Criteria:

* Participants with a history of the following diseases: cardiovascular, renal, hepatic, muscular, metabolic, gastrointestinal, neurologic, psychiatric, hematopoietic, respiratory, urinary, or other organic abnormalities as well as those participants who have had muscular trauma within 21 days previous to the study will also be excluded.
* Participants who require any kind of medication during the course of the study, apart from the IMP.
* Participants with a history of dyspepsia, gastritis, esophagitis, duodenal, or gastric ulcer, pyloro-duodenal obstruction, asthma, and urinary bladder obstruction.
* Participants with angle-closure glaucoma.
* Current or recent (within 14 days prior to administration of the IMP) use of monoamine oxidase inhibitors (MAOIs).
* Participants who have been exposed to enzyme or hepatic inducers or inhibitors within 30 days previous to the start of the study.
* Participants who have taken any type of medication including vitamin supplements (with or without prescription) or herbal remedies (e.g., St John's wort) within 30 days (or 7 half-lives) previous to the start of the study.
* Participants who have been hospitalized for any reason within 6 months prior to the start of the study.
* Participants who have taken IMPs from other investigations within 90 days prior to study start.
* Participants with a history of allergy or hypersensitivity to the study medication (doxylamine/pyridoxine), any other medication, food, or substance.
* Participants who have consumed alcohol, carbonated beverages and/or or beverages that contain methylxanthines (coffee, tea, cocoa, chocolate, mate, cola, etc.), grapefruit juice, or charbroiled foods within 12 hours prior to the start of the hospitalization period as well as participants who have smoked tobacco within 12 hours prior to the study start.
* Participants who have donated or lost more than 450 milliliters of blood within 60 days prior to study start.
* Current or recent use of depressants of the central nervous system such as alcohol.
* Participants with a history of dependence/abuse of alcohol, psychoactive substances or chronic use of medications.
* Participants requiring a special diet for any reason, e.g., vegetarian.
* Participants unable to understand the nature, objectives, and possible consequences of the study.
* Evidence of the participant's uncooperativeness during the conduct of the study.
* Participants with positive test results for drugs of abuse, pregnancy and/or alcohol in breath.
* Participants currently lactating.
* Participants receiving hormonal therapy via any route of administration.
* Participants who are not registered in the Comisión Federal para la Protección contra Riesgos Sanitarios (COFEPRIS) webpage.
* Relationship of subordination between the participants and the investigators.
* Sponsor or clinical site employees.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration curve from the administration until the time t (AUC0-t) of doxylamine | From pre-dose to 48 hours post-dose
  19 plasma samples will be collected from pre-dose to 48 hours post-dose. Doxylamine plasma concentrations will be determined using a high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay.
Maximum plasma concentration (Cmax) of doxylamine | From pre-dose to 48 hours post-dose
  19 plasma samples will be collected from pre-dose to 48 hours post-dose. Doxylamine plasma concentrations will be determined using a high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay.

SECONDARY OUTCOMES:
Area under the plasma concentration curve from 0 to infinity (AUC0-inf) of doxylamine | From pre-dose to 48 hours post-dose
  19 plasma samples will be collected from pre-dose to 48 hours post-dose. Doxylamine plasma concentrations will be determined using a high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay.
Time to maximum plasma concentration (Tmax) for doxylamine | From pre-dose to 48 hours post-dose
  19 plasma samples will be collected from pre-dose to 48 hours post-dose. Doxylamine plasma concentrations will be determined using a high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. Tmax will be calculated based on Cmax data for doxylamine.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Grünenthal GmbH

IPD SHARING:
Plan to Share IPD: No